CLINICAL TRIAL: NCT07332936
Title: Effect of Calcium Hydroxide vs. Tobradex Intracanal Medicament on Postoperative Endodontic Pain: A Prospective Trial
Brief Title: Tobradex as Intracanal Medicament
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Umm Al-Qura University (Other)
Responsible Party: Principal Investigator, Abdulaziz Bakhsh, Assistant Professor, Umm Al-Qura University
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: HAPO-02-K-012-2023-05-1631
Record Dates: First submitted 2025-12-30; First posted 2026-01-12 (Actual); Last update posted 2026-01-13 (Actual); Status verified 2026-01

CONDITIONS: Symptomatic Irreversible Pulpitis; Postoperative Endodontic Pain Following Emergency Root Canal Treatment
Keywords: Intracanal medication; Calcium Hydroxide; Tobradex; Pain; Root canal treatment
MeSH Terms: conditions — Pain | interventions — Calcium Hydroxide; Tobramycin, Dexamethasone Drug Combination

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tobramycin-Dexamethasone (Tobradex) (Experimental): Participants receive a tobramycin-dexamethasone combination (Tobradex) as an intracanal medicament following standardized emergency root canal treatment for symptomatic irreversible pulpitis.
  Interventions: Drug: Tobramycin + Dexamethasone
- Calcium Hydroxide (Active Comparator): Participants receive calcium hydroxide as an intracanal medicament following standardized emergency root canal treatment for symptomatic irreversible pulpitis.
  Interventions: Drug: Calcium Hydroxide (Ca(OH)2)

INTERVENTIONS:
Drug: Calcium Hydroxide (Ca(OH)2) — Calcium hydroxide is placed as an intracanal medicament after canal debridement during emergency root canal treatment as part of routine clinical practice.
  Arms: Calcium Hydroxide
Drug: Tobramycin + Dexamethasone — Tobramycin-dexamethasone (Tobradex) is placed as an intracanal medicament after canal debridement during emergency root canal treatment to reduce postoperative inflammation and pain.
  Arms: Tobramycin-Dexamethasone (Tobradex)

SUMMARY:
The goal of this prospective clinical study was to evaluate and compare the short-term effects of two intracanal medicaments-calcium hydroxide and a tobramycin-dexamethasone combination (Tobradex)-on postoperative pain following emergency root canal treatment in adult patients with symptomatic irreversible pulpitis.

The main question it aimed to answer was:

Does Tobradex reduce postoperative endodontic pain more effectively than calcium hydroxide within the first 48 hours after emergency root canal treatment? Adult patients presenting with acute dental pain and already receiving emergency root canal therapy as part of their routine clinical care were included. After canal debridement, patients received either calcium hydroxide or Tobradex as an intracanal medicament based on availability at the time of treatment. Participants reported their pain intensity using a numeric rating scale before treatment and again at 24 and 48 hours following the procedure. Pain outcomes were compared between groups, and the influence of demographic factors such as age and gender was also explored.

DETAILED DESCRIPTION:
This prospective clinical study investigates the effect of two commonly used intracanal medicaments-calcium hydroxide and a tobramycin-dexamethasone combination (Tobradex)-on postoperative pain following emergency root canal treatment. Postoperative pain remains a frequent concern after endodontic emergency procedures, particularly in teeth diagnosed with symptomatic irreversible pulpitis. While calcium hydroxide is widely used for its antimicrobial properties, evidence regarding its effectiveness in pain control is inconsistent. In contrast, intracanal medicaments containing corticosteroids have shown promise in reducing inflammation-related pain, yet limited clinical data are available for alternative steroid-antibiotic formulations such as Tobradex.

Patients presenting with acute endodontic pain and requiring emergency root canal treatment received standardized clinical care. Following canal debridement and irrigation, an intracanal medicament was placed, and the access cavity was temporized. The choice of medicament depended on availability during the emergency visit, reflecting real-world clinical practice. Pain intensity was assessed using a numeric rating scale at baseline and during the early postoperative period, allowing evaluation of both immediate and short-term pain reduction.

The primary focus of the study was to compare the magnitude and timing of pain relief achieved by the two medicaments within the first 48 hours after treatment. Secondary objectives included exploring whether patient-related factors, such as age or gender, influenced postoperative pain reduction. By examining pain outcomes during this critical early period, the study aims to clarify the potential benefit of incorporating a corticosteroid-antibiotic combination as an intracanal medicament in emergency endodontic care.

The findings of this study are intended to inform clinical decision-making regarding inter-appointment pain management and to provide preliminary evidence supporting alternative intracanal medicament strategies that prioritize patient comfort without compromising antimicrobial control.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 18 years or older
* Patients presenting with acute dental pain diagnosed as symptomatic irreversible pulpitis
* Teeth requiring emergency root canal treatment
* Ability to understand and provide informed consent
* Willingness to report pain levels during the follow-up period

Exclusion Criteria:

* Presence of acute or chronic apical abscess requiring systemic antibiotic therapy
* Teeth with previous root canal treatment
* Patients with systemic conditions that may affect healing or pain perception (e.g., uncontrolled diabetes, immunocompromised status)
* Known allergy or hypersensitivity to calcium hydroxide, tobramycin, dexamethasone, or related compounds
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-06-30 (Actual)

PRIMARY OUTCOMES:
Postoperative endodontic pain intensity | Baseline to 48 hours post-treatment
  Pain intensity measured using a numeric rating scale (0-10) at baseline, 24 hours, and 48 hours following intracanal medicament placement.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dental Medicine, Umm Al-Qura University, Mecca, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
Individual participant data collected during this study will not be shared publicly. Aggregate, de-identified results will be reported through publications and presentations.

REFERENCES:
- [Result] Alhilou AM, Al-Moraissi EA, Bakhsh A, Christidis N, Nasman P. Pain after emergency treatments of symptomatic irreversible pulpitis and symptomatic apical periodontitis in the permanent dentition: a systematic review of randomized clinical trials. Front Oral Health. 2023 Oct 18;4:1147884. doi: 10.3389/froh.2023.1147884. eCollection 2023. PMID 37920592